CLINICAL TRIAL: NCT03014440
Title: A Phase 1/2, Safety, Tolerability, and Dose-Finding Study of Cannabidiol for Drug-Resistant Epilepsies
Brief Title: Study of Cannabidiol for Drug-Resistant Epilepsies
Status: No longer available | Type: Expanded Access
Sponsor: Eric Marsh, MD (Other)
Collaborators: University of Pittsburgh (Other); Geisinger Clinic (Other)
Responsible Party: Sponsor-Investigator, Eric Marsh, MD, Assistant Professor of Pediatrics and Neurology, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Other Study IDs: 13-010562
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol
  Other Names: CBD; Epidiolex

SUMMARY:
The purpose of this study is to determine if cannabidiol is safe and effective at different doses as an additional treatment for pediatric drug-resistant epilepsy. Pure cannabidiol has potentially therapeutic properties, such as anti-convulsant effects, that may reduce seizure frequency. There are only a few open label studies that have demonstrated the safety and tolerance of cannabiodiol in both adult and pediatric epileptic populations--these studies were performed either retrospectively or with varying cannabidiol preparations. There are no well-documented studies and completely analyzed data for pediatric epileptic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 1 year old and 20 years old, male or female at the first visit, Week -4 (at time informed consent form is signed)
2. Documentation of a diagnosis of drug-resistant epilepsy as proven by and documented with medical records and/or the following clinical features (must have all 3 of the following):

   1. Failure to control seizures despite appropriate trial of 3 or more AEDs at therapeutic doses
   2. An intractable childhood epilepsy including, Dravet Syndrome or Lennox-Gastaut Syndrome
   3. Must report at least 3 countable (non-countable seizures includes absence and myoclonic) seizures per month
3. Between 1-3 baseline AEDs . Vagus nerve stimulator (VNS), ketogenic diet, and modified Atkins diet do not count towards this limit.
4. VNS must be on stable settings for a minimum of 3 months.
5. If on the ketogenic diet, must be on stable ratio for a minimum of 3 months.

Exclusion Criteria:

1. Epilepsies associated with neurodegenerative diseases, including neuronal ceroidolipofuscinosis, progressive myoclonus epilepsies, Rasmussen encephalitis, and tumors
2. Epilepsies associated with an inborn error of metabolism, including mitochondrial disorders
3. Felbatol initiated within the past 12 months
4. Use of any Cannabis-related product (including hemp oil) in the past 12 months as assessed by parental questioning.
5. Laboratory values on comprehensive metabolic panel (CMP) and complete blood count (CBC) testing that are Class 3 or higher according to the CTCAE v4.0.
6. Positive pregnancy test.

Ages: 1 Year to 20 Years | Sex: All
Age Groups: Child, Adult